CLINICAL TRIAL: NCT02077478
Title: Total Intravenous Anesthesia: TCI Versus MCI, Unresolved Question
Brief Title: Total Intravenous Anesthesia: TCI Versus MCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Riccardo Ragazzi, Associated professor, Università degli Studi di Ferrara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15022014
Record Dates: First submitted 2014-02-19; First posted 2014-03-04 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Test the Differences Between Schinder's TCI Model and MCI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MCI (Experimental): manually controlled infusion will be used
  Interventions: Device: Remifentanil and propofol administration using MCI
- TCI (Experimental): Target Controlled Infusion will be used
  Interventions: Device: Remifentanil and propofol administration using TCI

INTERVENTIONS:
Device: Remifentanil and propofol administration using TCI
  Arms: TCI
Device: Remifentanil and propofol administration using MCI
  Arms: MCI

SUMMARY:
test the following differences between Schinder's Target Controlled Infusion (TCI ) model and manually controlled infusion (MCI) :

* remifentanil and propofol total dose given
* incidence of awareness or inadequate anesthesia
* number of rescue dose given

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing breast or thyroid surgery

Exclusion Criteria:

* BMI > 35
* Surgery shorter than 30 minutes
* Patients with history of: alcol or drug abuse, kidney or liver failure, cardiovascular disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
incidence of awareness or inadequate anesthesia | every 3 minutes till the end of surgery

SECONDARY OUTCOMES:
remifentanil and propofol total dose given | every 30 minutes till the end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- 0532206570, Ferrara, Italy

REFERENCES:
- [Background] Russell D. Intravenous anaesthesia: manual infusion schemes versus TCI systems. Anaesthesia. 1998 Apr;53 Suppl 1:42-5. doi: 10.1111/j.1365-2044.1998.53s113.x. PMID 9640114